CLINICAL TRIAL: NCT01705210
Title: Functional MRI Biomarkers of Cognitive Decrements in Diabetes
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: NL34329.068.10 / METC 10-2-023; 916.11.059 (Other Grant/Funding Number: NWO/ZonMW VENI)
Record Dates: First submitted 2012-06-06; First posted 2012-10-12 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome X; Mild Cognitive Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diabetes mellitus type 2 (DM2)
- metabolic syndrome (MetS)
- healthy controls

SUMMARY:
The exact neuronal mechanism underlying the cognitive decline associated with diabetes mellitus type 2 (DM2) still remains to be elucidated. Multi-parametric functional MRI can potentially provide functional, micro-structural, micro-vascular, and metabolic information on the affected brain at an earlier stage than does conventional structural MRI. The overall aim of the current proposal is to obtain a better understanding in the neuronal mechanisms that underlie cognitive decline in DM2 and the putative prediabetic condition the metabolic syndrome (MetS).

DETAILED DESCRIPTION:
Diabetes mellitus type 2 (DM2) is a common chronic metabolic disorder that affects 4.1% of the Dutch population. In addition to vascular disease, DM2 is associated with structural brain changes visible on MRI, accelerated cognitive decline, and dementia in older individuals. The exact pathophysiological mechanisms underlying cognitive decrements in DM2 still remain to be elucidated. The 'metabolic syndrome' (MetS), defined as a cluster of cardiovascular risk factors (including obesity, hypertension, and dyslipidemia) is often considered a prediabetic condition. Individuals with MetS display similar cognitive decrements as do DM2 patients, but do not share the severity of brain injury. It has been indicated that in prediabetic MetS, cognitive problems precede structural brain changes, and that MetS and DM2 affect the brain through a shared mechanism in which vascular co-morbidity is essential.

The primary objectives are defined according to a hierarchical design: i) to tailor and apply multi-parametric, functional MRI techniques to identify cerebral abnormalities (cerebral biomarkers) in DM2 and MetS; ii) to investigate which cerebral biomarkers are shared and differ between DM2 and MetS; iii) to assess whether these cerebral biomarkers are associated with cognitive decrements.

ELIGIBILITY:
Inclusion criteria:

* Subjects aged 40-75 years
* Subjects enrolled in the existing 'Maastricht Study' (M-Study)
* Subjects gave written consent to be approached for additional research
* Subjects belongs to the 20% of the worst and 20% of the best performing (as based on neuropsychological cognitive testing (Stroop color-word test, 15 word learning test, and Delayed recall and recognition 15 word learning test)

Individuals Diabetes type 2:

- Fasting blood glucose ≥ 7.0 mmol/l, after an oral glucose tolerance test (OGTT)blood glucose ≥ 11.1 mmol/l or used oral glucose-lowering medication or insulin

Metabolic syndrome:

* Participants should meet three out of 5 of the following criteria [8]:

  1. Waist circumference > 88 cm (women), > 102 cm (men)
  2. Triglycerides ≥ 1.7 mmol/l
  3. HDL cholesterol < 1.3 mmol/l (women), < 1.0 mmol/l (men)
  4. Blood pressure ≥ 130/85 mmHg (or medication)
  5. Fasting blood glucose ≥ 6.1 mmol/l, after an OGTT blood glucose ≥ 7.8 mmol/l

     Control participants:
* Those who fulfilled no more than 1 criterium of the metabolic syndrome, no DM2.

Exclusion criteria:

* Contra-indications for MRI examination (e.g. pacemaker; neurostimulator; medication pump; cochlear or hearing implant; tattoos or other items that cannot be removed and include metal parts (for instance from operations in the past); metal splinter in the eye; pregnancy and claustrophobia; brain vessel clamps; denture, which contains magnets).
* Psychiatric co-morbidity and inability to perform the functional MRI tests.
* Incomplete cognitive assessment data
* Diabetes mellitus type 1 (DM1)
* Subjects who are not belonging to the 20% of the worst and 20% of the best performing individuals (as based on neuropsychological cognitive testing (Stroop color-word test, 15 word learning test, and Delayed recall and recognition 15 word learning test).
* Last visit of the subjects to the M-Study should be less than one year

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Matched subjects aged 40-75 years with Diabetes mellitus type 2, metabolic syndrome, and healthy controls
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2012-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Functional and structural connectivity relationships of multiple brain regions and biomarkers of brain alterations | subjects will be assessed once (on 1 day)
  Differences in macro-structural, micro-structural, and metabolic concentrations between patients and healthy controls will be evaluated. These MRI measures include volumetric characteristics (e.g. hyper-intensities, white matter lesions, atrophy), quantitative measures (e.g. T2 relaxation times, mean diffusivity, fractional anisotropy), functional characteristics (e.g. activated regions, cerebral blood flow), metabolic characteristics (e.g. concentration of metabolites), network properties (e.g. functional and structural connectivity, graph-theoretical measures).

SECONDARY OUTCOMES:
Anthropometrics | subjects will be assessed once (on 1 day)
  Simple anthropometric measurements will include: Body mass index will be calculated as the weight (kg) divided by the square of the height (m). Waist circumference (WC) will be taken as the minimum circumference between the umbilicus and xiphoid process and measured to the nearest 0.5 cm.
Mental health | subjects will be assessed once (on 1 day)
  For assessment of mental health, specifically depression, the Cambridge Mental Disorders of the Elderly Examination will be used.
Lifestyle | subjects will be assessed once (on 1 day)
  Lifestyle specifics, including alcohol consumption, smoking behavior and mobility will be obtained through a questionnaire.
Cardiovascular risk factors | subjects will be assessed once (on 1 day)
  Blood samples will be assessed for:
  Fasting circulating levels of glucose, albumin, creatinin, total cholesterol, LDL- and HDL-cholesterol, triglycerides, HbA1c and uric acid.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus FA Jansen, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Result] van Bussel FC, Backes WH, Hofman PA, van Oostenbrugge RJ, Kessels AG, van Boxtel MP, Schram MT, Stehouwer CD, Wildberger JE, Jansen JF. On the interplay of microvasculature, parenchyma, and memory in type 2 diabetes. Diabetes Care. 2015 May;38(5):876-82. doi: 10.2337/dc14-2043. Epub 2015 Feb 17. PMID 25690006